CLINICAL TRIAL: NCT05705219
Title: Development of 3D Multi-Parametric Ultrasound (MPUS) as a Decision Support Tool for Patients With Abdominal and Pelvic Tumors Undergoing Therapy
Brief Title: Development of 3D Multi-Parametric Ultrasound (MPUS) as a Decision Support Tool for Patients
Acronym: 3DMPUS
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ahmed El Kaffas, Associate Professor, University of California, San Diego
Other Study IDs: IRB-68310; R01CA195443 (NIH); NCI-2024-03676 (Other: CTRP)
Record Dates: First submitted 2023-01-18; First posted 2023-01-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Liver Cancer, Adult
Keywords: Diagnostic Study
MeSH Terms: conditions — Carcinoma, Hepatocellular; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- 3-dimensional multi-parametric ultrasound imaging (3D-MPUS): Participants will receive sulfur hexafluoride IV and undergo 3D-MPUS imaging over 20 minutes.
  Interventions: Diagnostic Test: 3D-MPUS

INTERVENTIONS:
Diagnostic Test: 3D-MPUS — Participants will receive approximately < 20 minutes ultrasound scan to locate the lesion followed by acquisition of 3D-MPUS acquisition.
  Other Names: 3-dimensional multi-parametric ultrasound imaging

SUMMARY:
This clinical trial studies how well 3-dimensional multi-parametric ultrasound (3D MPUS) imaging works as a decision-support tool for patients with liver tumors undergoing therapy. Continuous and dynamic imaging of patients undergoing therapy is required to monitor early-phase treatment response.

DETAILED DESCRIPTION:
This clinical trial studies how well 3-dimensional multi-parametric ultrasound (3D MPUS) imaging works as a decision-support tool for patients with liver tumors undergoing therapy. Continuous and dynamic imaging of patients undergoing therapy is required to monitor early-phase treatment response. 3D-MPUS is an inexpensive and safe method, which may provide complementary quantitative functional (perfusion) and tissue characterization information to anatomical radiological assessment or blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has untreated liver metastases from colorectal low-grade adenocarcinoma (biopsy-proven and/or characteristic findings on CT, MRI, or FDG-PET) and has planned to undergo a new course of cancer therapy*.
2. Participant is age >/=18 years.
3. Participant has at least one target lesion that measures ≥1cm in diameter (minimum size according to RECIST 1.1) with a maximum diameter of 14cm amenable to imaging with ultrasound
4. Participant is willing to comply with protocol requirements.
5. Participant has given written informed consent to participate in this study.

   * Any line of cancer therapy is allowed, including systemic and localized treatments, after any prior treatment. For systemic combination treatments, prior treatment with either drug is allowed at the discretion of the investigators, including rechallenges with the same drug combination, for example upon progression on imaging after a treatment break. For combination treatments where patients start treatment with different drugs at different times, the start date of treatment is determined at the discretion of the investigators and can be the start date of the first drug or of the combination treatment. Repeat participation in the study is allowed, if patients are eligible again per their treatment plan.

Exclusion Criteria:

1. Participant has documented anaphylactic or other severe reaction to any ultrasound contrast media or polyethylene glycol (PEG).
2. Participant has any comorbid condition** that, in the opinion of the treating provider or the Protocol Director, compromises the participant's ability to participate in the study.
3. Participant is pregnant (positive urine or serum beta-hCG) or lactating.
4. Presence of cardiac shunt or presence of pulmonary hypertension (contradiction for ultrasound contrast agent)
5. Renal insufficiency with a creatinine level >1.5mg/dl, per our institutional guidelines (contradiction for CT imaging).

   * Examples: any mental condition that compromises the ability to follow a consent discussion, or to make informed decisions (except if represented by a Legally Authorized Representative [LAR]); any condition that makes the participant not a good candidate to have ultrasound exams with contrast agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. The participant is about to undergo a new course of therapy for primary or metastatic cancer in the abdominal or pelvic region.
  2. The participant is age > 18 years.
  3. Participant has at least one target lesion (≥1cm and <14cm)
  4. The participant is willing to comply with protocol requirements.
  5. The participant has the ability to understand and the willingness to sign a written informed consent document.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of the 3D-MPUS data acquisition | Baseline visit
  Diagnostic yield will be the percentage of non-missing measurements (per reader, per measurement)
  Participants with successful measurements of the following parameters (following administration of a contrast agent).
  * peak enhancement (PE)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El Kaffas, PhD, Principal Investigator — University of California, San Diego; Aya Kamaya, MD, Study Director — Stanford University; Andrej Lyshchik, MD, PhD, Study Director — Thomas Jefferson University; Aman Khurana, MD, Study Director — University of California, San Diego; Yuko Kono, MD, PhD, FAIUM, FAASLD, Study Director — University of California, San Diego
Locations (3):
- United States (3):
  - Stanford University, School of Medicine, Palo Alto, California
  - University of California, San Diego, San Diego, California
  - Thomas Jefferson Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No